CLINICAL TRIAL: NCT00161486
Title: The Effects of Testosterone on Prostate Tissue in Normal Men (ACYP-1)
Brief Title: The Effects of Testosterone on Prostate Tissue (ACYP-1)
Acronym: ACYP-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: William J Bremner, MD, PhD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-9401-B; U 54 HD42454
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Hypogonadism; Contraception
Keywords: Male contraception; Prostate; Acyline; Androgen replacement
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; acyline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo acyline injections every two weeks (2 doses) + placebo testosterone gel daily for 4 weeks
  Interventions: Drug: Placebo acyline; Drug: Placebo Testosterone gel
- 2 (Active Comparator): Acyline 300 μg/kg every two weeks (2 doses) + placebo Testosterone gel daily for 4 weeks
  Interventions: Drug: Acyline; Drug: Placebo Testosterone gel
- 3 (Active Comparator): Acyline 300 μg/kg every two weeks (2 doses) for 4 weeks + Testosterone gel 100 mg daily for 4 weeks
  Interventions: Drug: Testosterone gel; Drug: Acyline

INTERVENTIONS:
Drug: Testosterone gel — Testosterone gel 100 mg daily for 4 weeks
  Other Names: Testim
  Arms: 3
Drug: Acyline — Acyline 300 μg/kg every two weeks (2 doses) for 4 weeks
  Arms: 2; 3
Drug: Placebo acyline — Placebo acyline injections every two weeks (2 doses)
  Arms: 1
Drug: Placebo Testosterone gel — placebo testosterone gel daily for 4 weeks
  Arms: 1; 2

SUMMARY:
The purpose of this research study is to understand the effects of testosterone on the prostate. This knowledge will be used to help in the development of a safe male hormonal contraceptive and may impact the development of androgen replacement therapy in older men.

DETAILED DESCRIPTION:
We will be administering two drugs: Testim (testosterone gel) and Acyline. Acyline is an experimental drug. We want to see their effects on levels of hormones in the blood and prostate. In addition, we will be examining the effects of these drugs on the expression of genes within the prostate.

Acyline suppresses LH and FSH, which are hormones made by the pituitary gland, thus blocking the signal from the brain that causes the testes to make testosterone. Therefore, Acyline blocks testosterone production. In preliminary studies, a single injection of Acyline reversibly lowered the FSH, LH and testosterone levels in the blood for approximately 15 days. Prolonged low levels of LH and FSH cause suppression of sperm production in normal men. However, men may experience some side effects from the low levels of testosterone caused by acyline, thus exogenous testosterone is required to sustain normal male androgen and organ effects without suppressing spermatogenesis. This combination of drugs is a promising male contraceptive regimen. In addition, millions of older men are using testosterone replacement to treat male "andropause"; low level testosterone associated with aging. However, the effect of testosterone on the prostate is unknown. Studies examining the effect of testosterone on the prostate are needed.

ELIGIBILITY:
Inclusion Criteria:

* Males between 35 and 55, normal serum testosterone levels, normal gonadal function

Exclusion Criteria:

* History of prostate cancer, PSA>2.0, AUA BPH symptom score >10, History of testosterone or anabolic steroid use, chronic medical illness or prostate disease, active serious infection or immunosuppression, history of a bleeding disorder or need for anticoagulation, abnormal digital rectal exam, abnormal prostate ultrasound, first degree relative with history of prostate cancer

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2004-07; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Intervention trial to examine the hormonal regulation of prostate gene expression and tissue hormone levels, tissue protein expression and apoptosis. | 28-days

SECONDARY OUTCOMES:
Cellular immune function | 28-days

CONTACTS AND LOCATIONS:
Overall Officials: William J Bremner, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Bhasin S, Singh AB, Mac RP, Carter B, Lee MI, Cunningham GR. Managing the risks of prostate disease during testosterone replacement therapy in older men: recommendations for a standardized monitoring plan. J Androl. 2003 May-Jun;24(3):299-311. doi: 10.1002/j.1939-4640.2003.tb02676.x. No abstract available. PMID 12721204
- [Background] Morgentaler A, Bruning CO 3rd, DeWolf WC. Occult prostate cancer in men with low serum testosterone levels. JAMA. 1996 Dec 18;276(23):1904-6. PMID 8968017
- [Background] Schatzl G, Madersbacher S, Thurridl T, Waldmuller J, Kramer G, Haitel A, Marberger M. High-grade prostate cancer is associated with low serum testosterone levels. Prostate. 2001 Apr;47(1):52-8. doi: 10.1002/pros.1046. PMID 11304729
- [Background] Nelson PS, Clegg N, Arnold H, Ferguson C, Bonham M, White J, Hood L, Lin B. The program of androgen-responsive genes in neoplastic prostate epithelium. Proc Natl Acad Sci U S A. 2002 Sep 3;99(18):11890-5. doi: 10.1073/pnas.182376299. Epub 2002 Aug 16. PMID 12185249
- [Background] Herbst KL, Anawalt BD, Amory JK, Bremner WJ. Acyline: the first study in humans of a potent, new gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2002 Jul;87(7):3215-20. doi: 10.1210/jcem.87.7.8675. PMID 12107227
- [Background] Bagatell CJ, Matsumoto AM, Christensen RB, Rivier JE, Bremner WJ. Comparison of a gonadotropin releasing-hormone antagonist plus testosterone (T) versus T alone as potential male contraceptive regimens. J Clin Endocrinol Metab. 1993 Aug;77(2):427-32. doi: 10.1210/jcem.77.2.8345047.
- [Background] Swerdloff RS, Bagatell CJ, Wang C, Anawalt BD, Berman N, Steiner B, Bremner WJ. Suppression of spermatogenesis in man induced by Nal-Glu gonadotropin releasing hormone antagonist and testosterone enanthate (TE) is maintained by TE alone. J Clin Endocrinol Metab. 1998 Oct;83(10):3527-33. doi: 10.1210/jcem.83.10.5184. PMID 9768659
- [Background] Tom L, Bhasin S, Salameh W, Steiner B, Peterson M, Sokol RZ, Rivier J, Vale W, Swerdloff RS. Induction of azoospermia in normal men with combined Nal-Glu gonadotropin-releasing hormone antagonist and testosterone enanthate. J Clin Endocrinol Metab. 1992 Aug;75(2):476-83. doi: 10.1210/jcem.75.2.1639948.
- [Result] Page ST, Plymate SR, Bremner WJ, Matsumoto AM, Hess DL, Lin DW, Amory JK, Nelson PS, Wu JD. Effect of medical castration on CD4+ CD25+ T cells, CD8+ T cell IFN-gamma expression, and NK cells: a physiological role for testosterone and/or its metabolites. Am J Physiol Endocrinol Metab. 2006 May;290(5):E856-63. doi: 10.1152/ajpendo.00484.2005. Epub 2005 Dec 13. PMID 16352669
- [Result] Page ST, Lin DW, Mostaghel EA, Hess DL, True LD, Amory JK, Nelson PS, Matsumoto AM, Bremner WJ. Persistent intraprostatic androgen concentrations after medical castration in healthy men. J Clin Endocrinol Metab. 2006 Oct;91(10):3850-6. doi: 10.1210/jc.2006-0968. Epub 2006 Aug 1. PMID 16882745
- [Result] Mostaghel EA, Page ST, Lin DW, Fazli L, Coleman IM, True LD, Knudsen B, Hess DL, Nelson CC, Matsumoto AM, Bremner WJ, Gleave ME, Nelson PS. Intraprostatic androgens and androgen-regulated gene expression persist after testosterone suppression: therapeutic implications for castration-resistant prostate cancer. Cancer Res. 2007 May 15;67(10):5033-41. doi: 10.1158/0008-5472.CAN-06-3332. PMID 17510436